CLINICAL TRIAL: NCT02833402
Title: The Association Between the Urinary Microbiome and Response to Sacral Neuromodulation in Women With Urgency Urinary Incontinence
Brief Title: Sacral Neuromodulation and the Microbiome
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: American Urogynecologic Society (Other); University of Pennsylvania (Other); University of Missouri-Columbia (Other); University of North Carolina (Other); University of Washington (Other); Saint Francis Hospital and Medical Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: STU00202669
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Urgency Urinary Incontinence
Keywords: Sacral Neuromodulation; Urinary leakage; Urinary incontinence; Urinary microbiome
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will be obtaining urine specimens for microbial analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UUI patients undergoing SNM: Urine specimens, questionnaire, and medical data will be collected from subjects that have UUI and are undergoing InterStim placement (SNM).
  Interventions: Device: InterStim Therapy

INTERVENTIONS:
Device: InterStim Therapy — Sacral Neuromodulation, delivered by the InterStim® System, offers long-term control of bladder control and bowel control symptoms through modulation of the nerves that help control the pelvic floor and lower urinary tract.
  Other Names: Sacral Neuromodulation

SUMMARY:
Sacral neuromodulation (SNM) which is approved as a treatment for men and women with urgency urinary incontinence (UUI), urgency frequency syndrome, urinary retention and anal incontinence, is a procedure designed to deliver electrical pulses to the sacral nerves, thereby influencing the bladder, sphincters, and pelvic floor. Although the success rates of this treatment are quite high, the precise mechanism of action of SNM in subjects with UUI remains unclear. Moreover, there are little data regarding specific patient characteristics that may serve as "predictors" for SNM success. Recent studies suggest that the bacterial community that lives in the urinary tract plays a role in the development and continuation of urinary symptoms. It is proposed that the urinary microbiome may change in women before and after SNM implantation and this study aims to describe these changes. Investigators in this study also hope to determine if differences in the urinary microbiome exist in women with a positive response to SNM treatment (responders) compared to those without symptom improvement (non-responders). This hypothesis will be tested by collecting urine samples as well as questionnaire and medical data from subjects with UUI that are already planning on undergoing SNM as part of clinical care before and after their SNM treatment.

DETAILED DESCRIPTION:
One in four women reports bothersome symptoms of a pelvic floor disorder with 16% reporting urinary incontinence (UI). Sacral neuromodulation (SNM) which is approved for men and women with urgency urinary incontinence (UUI), urgency frequency syndrome, urinary retention and anal incontinence, is a procedure designed to deliver electrical pulses to the sacral nerves, thereby influencing the bladder, sphincters, and pelvic floor. SNM provides symptomatic relief in 70-86% of patients undergoing the procedure for UUI according to several recent prospective studies. Although the success rates are quite high, the precise mechanism of action of SNM in subjects with UUI remains unclear. Moreover, there are little data regarding specific patient characteristics that may serve as "predictors" for SNM success.

The microbiome refers to the genetic material of the micro-organisms present in a particular environment. The role of the microbiome has recently been implicated in several disease states (obesity, inflammatory bowel disease, and functional bowel disease. Initially, the urinary microbiome was not a part of the "human microbiome project" as it was widely accepted that urine is sterile. However, recent studies have noted the presence of a urinary microbiota in adult women without clinical urinary tract infections. Furthermore, recent studies have shown that the urinary microbiome differs among women with UUI versus those without UUI and also among women with interstitial cystitis / painful bladder syndrome versus those without it. These studies suggest that the urinary microbiome plays a role in the development and continuation of urinary symptoms.

Because of the invasiveness of the SNM procedure, it would be helpful to have a way to predict treatment success. Investigators in this study propose that the urinary microbiome may change in women before and after SNM implantation and hope to describe these changes by conducting this study. Investigators also hope to determine if differences in the urinary microbiome exist in women with a positive response to SNM treatment (responders) compared to those without symptom improvement (non-responders). This hypothesis will be tested by collecting urine samples from subjects with UUI that are already planning on undergoing SNM as part of clinical care before and after their SNM treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 with UUI planning to undergo SNM implantation will be included if they have at least 2 UUI episodes on a baseline 3-day diary.
* Willing and able to complete study visits, questionnaires and diaries
* Women previously treated with OAB medication are permitted to participate, but must be off of all medications for a minimum of 4 weeks prior to the performance of the baseline 3-day bladder diary and baseline assessments. They will be required to stay off any OAB medications for the duration of the study.

Exclusion Criteria:

* Neurologic disease (including multiple sclerosis, spinal cord injury, history of cerebrovascular accident, significant peripheral neuropathy)
* Pregnancy
* History of recurrent UTI in last 6 months by definition (3 culture proven UTI in 1 year or 2 culture proven UTI in 6 month period), or women who are receiving treatment for recurrent UTI
* Prolapse beyond the hymen
* Other contraindication to SNM
* Microscopic hematuria, as defined as 3 or more RBC/hpf on complete microscopic urinary analysis, without appropriate work-up (renal imaging and cystoscopy)
* History of pelvic radiation
* History of previous neuromodulation therapy including intravesical botulinum toxin, sacral neuromodulation or peripheral tibial nerve stimulation.

Deferral Criteria:

* Recent systemic antibiotic exposure (within the past 4 weeks)
* Urinary Tract Infection (UTI) at time of enrollment or sample

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women over the age of 18 with UUI planning to undergo placement of a sacral nerve modulator will be included if they have at least 2 UUI episodes on a 3-day diary.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
The abundance of bacteria associated with inflammatory processes in the urinary tract of women with a positive response to SNM (responders) versus those without symptom improvement (non-responders) | 3 months after SNM treatment treatment

SECONDARY OUTCOMES:
Changes in the urinary microbial community of responders to SNM therapy | 3 months after initiating SNM treatment

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Mueller, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No